CLINICAL TRIAL: NCT05529706
Title: Community-based Brain Health Program to Address Dementia Risk
Acronym: C-BBHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: YMCA of San Francisco (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-0318-22
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Health Program (Experimental): A multimodal educational and interactive diet, exercise and computerized cognitive exercise public health program.
  Interventions: Other: Brain Health Program

INTERVENTIONS:
Other: Brain Health Program — The Brain Health Program employs 1-hour/week group-based training and education regarding modifiable Alzheimer's disease dementia risk factors delivered over a 12-week period. Participants will be assigned into a group of up to 20 participants, and participants will engage the Brain Health Program collaboratively, as administered by the program content leader (instructor), while also being monitored and supported by the tech leader (in accordance with the Diabetes Prevention Program model).

SUMMARY:
This is a validation study to evaluate the acceptability, feasibility and preliminary efficacy of the Brain Health Program, a multimodal curriculum covering dementia risk factors and evidence-based change interventions. The goal of this study is to evaluate the Brain Health Program in individuals with identified risk factors for the onset of dementia and to prepare for a large-scale efficacy trial in this population.

DETAILED DESCRIPTION:
This study will employ an evidence-based Brain Health Program curriculum, which involves a twelve-week, group-administered, personalized program designed to improve brain health in individuals with identified risk factors for the onset of dementia. This is a single-arm open-label feasibility study, enrolling older adults with Alzheimer's disease risk factors in a public health, community-deployed, group-based and individualized multimodal Brain Health Program (targeting, among other domains, diet, exercise and cognitive exercise), with a set of baseline assessments intended to characterize the population, and outcome measure to evaluate the usability of the program, as well as preliminary efficacy to reduce dementia risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 65 years of age or older.
2. Participants who meet criteria for one or more ADRD dementia risk factors

   1. Family history of Alzheimer's dementia (1st degree relative)
   2. Genetic marker (APOE4++)
   3. Subjective or objective cognitive decline (neuropsychological testing; or self-reported "yes" to the following question: "In the past two years, have you experienced a decline in your memory or thinking?"
   4. Poorly controlled hypertension or diabetes
   5. Physical inactivity <150min/week per Surgeon General guidelines
   6. Social isolation, in which participant rarely or never gets social and emotional support when needed
3. Participants who are fluent English or Spanish speakers, per self-report, to ensure reasonable neuropsychological results on key assessments.
4. Participants have access to an internet accessible device (eg. laptop, desktop computer, tablet or smartphone)
5. Participants are able to attend all 12 classes (once a week for 12 weeks) and make up missed classes, as needed
6. Participants are able to travel to/from YMCA location, if they choose to be a part of the in-person group

Exclusion Criteria:

1. Inability to provide informed consent
2. Cognitive Abilities Screening Instrument - Short (CASI-Short) scores ≤ 25 (suggestive of cognitive impairment)
3. Participants with untreated psychiatric conditions, including substance abuse/dependence disorders.
4. Participants enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment that could affect the outcome of this study. However, participation in standard treatments (e.g., occupational therapy) or use of prescribed medications (e.g., anti-depressants) is allowable.
5. Participants presently attending classes or courses like this program that is focused on dementia risk and behavior management.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Net Promoter Score | At 12 weeks
  The scoring for this answer is based on a 0 to 10 scale. Those who respond with a score of 9 to 10 are called Promoters, and are considered likely to exhibit value-creating behaviors, such as making more positive referrals to other potential program participants. Those who respond with a score of 0 to 6 are labeled Detractors, and they are believed to be less likely to exhibit the value-creating behaviors. Responses of 7 and 8 are labeled Passives, and their behavior falls between Promoters and Detractors. The Net Promoter Score is calculated by subtracting the percentage of customers who are Detractors from the percentage of customers who are Promoters. For purposes of calculating a Net Promoter Score, Passives count toward the total number of respondents, thus decreasing the percentage of detractors and promoters and pushing the net score toward 0.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- YMCA of San Francisco, San Francisco, California, United States